CLINICAL TRIAL: NCT00004826
Title: Study of Clozapine for the Treatment of Psychosis in Patients With Idiopathic Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Hospital of Rhode Island (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13295; MHRI-FDR001416
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1998-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Parkinson Disease; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Clozapine

INTERVENTIONS:
Drug: clozapine

SUMMARY:
OBJECTIVES: I. Determine the efficacy and tolerability of clozapine in ameliorating psychosis in patients with idiopathic Parkinson's disease (PD).

II. Determine the adverse effects of clozapine on motor function in this patient population.

III. Determine the safety of clozapine in psychotic PD patients taking multiple anti-PD medications.

IV. Describe the phenomenology of drug induced psychosis in PD.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, placebo controlled, double blind study, followed by an open label treatment of all patients. Patients are stratified according to the institutional investigator and age.

In the first phase of the study, patients receive either clozapine or placebo. The drug is taken orally at night, approximately 30 minutes before retiring. Therapy continues for 4 weeks unless psychosis becomes unmanageable without hospitalization, parkinsonism worsens, or other adverse effects occur. It is possible that the dose may be escalated.

In the second phase of the study, all patients are treated with open label clozapine. Therapy continues for 3 months unless psychiatric status or parkinsonism progress. Dose escalation is also possible during this phase.

Patients are followed weekly during the first phase of the study, and monthly during the second phase.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Presumed idiopathic Parkinson's disease Presence of three of the cardinal features: Rest tremor Rigidity Bradykinesias/akinesia Postural and balance abnormalities Absence of alternative explanations for the syndrome Absence of atypical features Psychosis of at least 4 weeks duration requiring treatment --Prior/Concurrent Therapy-- Chemotherapy: No concurrent chemotherapy Other: No use of any dopamine blocking drug within the past 3 months No use of depot neuroleptic within the past 12 months No change of antidepressant or anxiolytic dose within the past 1 month No prior clozapine for psychosis Anti-PD medications stable for at least 7 days before study entry --Patient Characteristics-- Hematopoietic: No history of leukopenia No active blood dyscrasia other than mild anemia Renal: No active problems with urinary retention Cardiovascular: No symptomatic orthostatic hypotension No uncontrolled angina No myocardial infarction within the past 3 months Other: Fertile patients must use effective contraception No uncontrolled seizures (i.e., 1 or more seizures per month over the past 6 months) No dementia precluding accurate assessment on psychiatric assessment battery No AIDS No other illness that would make use of clozapine potentially hazardous No narrow angle glaucoma No systemic factor contributing to the psychosis (e.g., urinary infection, liver disease, renal failure, anemia, infection, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 1993-10; Study Completion 1997-11

CONTACTS AND LOCATIONS:
Overall Officials: Joseph H. Friedman, Study Chair — Memorial Hospital of Rhode Island